CLINICAL TRIAL: NCT01633892
Title: Use of Concentrated Endogenous Autologous Adipose Stromal Cells in Fat Grafts for Craniofacial Trauma
Acronym: ARM5
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding ended
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, J. Peter Rubin, MD, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO12010078
Record Dates: First submitted 2012-06-21; First posted 2012-07-04 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-04

CONDITIONS: Craniofacial Injuries
Keywords: Craniomaxillofacial (CMF); Battle-injured (BI); Facial Trauma; Fat Grafts; Autogenous Fat Transfers (AFT); Wounded warriors; Adipose Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fat Grafting (Experimental)
  Interventions: Procedure: Fat Grafting

INTERVENTIONS:
Procedure: Fat Grafting

SUMMARY:
Traumatic facial injuries, especially those sustained in military combat, are characterized by destruction of bone and soft tissue. While the bony structures of the face can be reconstructed, it is difficult to return the soft tissue back to its original form. Many times, fat grafting, a common cosmetic and reconstructive procedure, is used in hopes of improving the soft tissue deformity. Fat grafting is a procedure in which a person's own fat is taken from areas throughout the body, usually the thighs or abdomen, with a small liposuction tube. The fat is then transferred into the area that has lost volume or fullness. The fullness of the soft tissue area may decrease over time because the transferred fat can be reabsorbed by the body. Altering the current fat grafting procedure, slightly, could lead to less reabsorption and a lasting fullness of the soft tissue area outcome of the fat graft procedure.

The investigators are conducting this research study to help us improve the surgical treatment of people who have suffered facial soft tissue loss as a result of trauma. The goal of this research study is to see how each person's fat grafts will maintain the fat over time and to measure the quality of life during a 9 month post-surgical follow-up period. The total duration of participation is approximately 11-12 months. In this study, the investigators will concentrate the fat in the fat grafting procedure to determine whether this process will maintain the fat over time. The areas treated with enhanced fat grafts will be compared with areas treated with standard of care fat grafts. At least two areas of your face will be treated with fat grafts, (standard of care fat grafts and concentrated fat grafts).

This study is the second of two clinical studies at the University of Pittsburgh using each person's fat graft with concentration of fat cells in the graft to observe if there is less fat resorption compared to using fat grafts alone. Each study is using a different concentration of fat in the fat graft compared to the first clinical study.

DETAILED DESCRIPTION:
Craniofacial injuries have serious psychosocial sequele and affect quality of life. Many individuals who suffer significant facial disfigurement from injury experience psychological distress and impairment in functioning not limited to the acute phase of injury, but over a longer term period of treatment, recovery, and adjustment. Until recently, treatment of disfiguring craniofacial injuries has been mostly limited to surgical flap procedures, microsurgical tissue transfer, and implantable prostheses. However, these methods can leave conspicuous scars on the face and the donor site, and in the case of implants can lead to complications associated with foreign materials. Autologous fat grafting with minimally invasive cannulas is a procedure that has been used for decades in common plastic surgery practice for facial aesthetic procedures. This technique is also a promising treatment for soft tissue reconstruction after craniofacial trauma because the graft harvest and injection are minimally invasive. The treatment is performed by using a small liposuction cannula to aspirate fat tissue from the donor site, and then re-injecting the fat into the recipient site with specialized injection cannulas. After harvest, and prior to injection, the fat graft is subjected to a mechanical processing step to separate the aqueous layer and concentrate the adipocytes. This often takes the form of centrifugation or filtering.

The main problem with autologous fat grafting is a variable resorption of the graft volume over time. As much as 30-60% of the graft volume can diminish over time. Many variables may influence the behavior of clinical fat grafts, including harvest site, harvest technique, graft preparation, and injection technique.

Concentrating the already present autologous adipose stromal cells within the fat grafts is not expected to increase subject risk levels beyond the risk levels of the application of fat grafts. We are currently approved for the application of fat grafts with concentrated autologous adipose stromal cells [IRB#10100293]. This proposal uses an increased concentration of adipose stromal cells compared to the above referenced study; no increase of risk to the subject is anticipated. We hypothesize that fat grafting for facial trauma, facilitated by enhancing graft quality with a higher concentration of endogenous autologous vascular adipose stromal cells in the grafted tissue, will enhance the successful restoration of tissue volume and craniofacial form. The use of a higher concentration of autologous adipose stromal cells may lead to lower fat resorption rates that may be observed in the approved IRB study [PRO10100293]. Additionally, we hypothesize that the clinical results using the concentrated autologous stromal vascular cells will be durable and the subject's quality of life scores will be improved compared to subjects who have had fat grafting alone using historical controls.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older and able to provide informed consent.
2. Have suffered injury resulting in craniofacial volume defects which could be treated with a graft volume of between 3 and 100 cc of lipoaspirate
3. Be at least 3 months post-injury or post-surgery (from trauma procedures) so that acute edema is resolved
4. Volume defects are covered by intact skin and do not communicate with oral cavity or sinuses
5. The three dimensional geometry of the volume defects would allow for treatment with lipoaspirate injection so that at least two distinct treated areas could be discerned on gross examination and radiographically (e.g. treated regions are on opposite sides of the face, on lower face versus upper face, or separated by a bony landmark such as zygoma. This would include the ability to treat an uninjured regions with fat grafts in order to obtain symmetry or balance.
6. Willing and able to comply with follow up examinations,

Exclusion Criteria:

1. Age less than 18 years
2. Inability to provide informed consent
3. Craniofacial defects intended for treatment have open wounds or communicate with oral cavity or sinus (note: presence of such a defect in the setting of another defect(s) that meets treatment criteria will not exclude the patient from participating).
4. Active infection anywhere in the body
5. Diagnosed with cancer within the last 12 months and/or presently receiving chemotherapy or radiation treatment
6. Known coagulopathy
7. Systemic disease that would render the fat harvest and injection procedure, along with associated anesthesia, unsafe to the patient.
8. Pregnancy
9. Diagnosis of Schizophrenia or Bipolar Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Peter Rubin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yoshimura K, Sato K, Aoi N, Kurita M, Hirohi T, Harii K. Cell-assisted lipotransfer for cosmetic breast augmentation: supportive use of adipose-derived stem/stromal cells. Aesthetic Plast Surg. 2008 Jan;32(1):48-55; discussion 56-7. doi: 10.1007/s00266-007-9019-4. Epub 2007 Sep 1. PMID 17763894
- [Background] Masuda T, Furue M, Matsuda T. Novel strategy for soft tissue augmentation based on transplantation of fragmented omentum and preadipocytes. Tissue Eng. 2004 Nov-Dec;10(11-12):1672-83. doi: 10.1089/ten.2004.10.1672. PMID 15684676
- [Background] Matsumoto D, Sato K, Gonda K, Takaki Y, Shigeura T, Sato T, Aiba-Kojima E, Iizuka F, Inoue K, Suga H, Yoshimura K. Cell-assisted lipotransfer: supportive use of human adipose-derived cells for soft tissue augmentation with lipoinjection. Tissue Eng. 2006 Dec;12(12):3375-82. doi: 10.1089/ten.2006.12.3375. PMID 17518674
- [Background] Moseley TA, Zhu M, Hedrick MH. Adipose-derived stem and progenitor cells as fillers in plastic and reconstructive surgery. Plast Reconstr Surg. 2006 Sep;118(3 Suppl):121S-128S. doi: 10.1097/01.prs.0000234609.74811.2e. PMID 16936551
- [Background] Lu F, Li J, Gao J, Ogawa R, Ou C, Yang B, Fu B. Improvement of the survival of human autologous fat transplantation by using VEGF-transfected adipose-derived stem cells. Plast Reconstr Surg. 2009 Nov;124(5):1437-1446. doi: 10.1097/PRS.0b013e3181babbb6. PMID 20009828
- [Background] Zhu M, Zhou Z, Chen Y, Schreiber R, Ransom JT, Fraser JK, Hedrick MH, Pinkernell K, Kuo HC. Supplementation of fat grafts with adipose-derived regenerative cells improves long-term graft retention. Ann Plast Surg. 2010 Feb;64(2):222-8. doi: 10.1097/SAP.0b013e31819ae05c. PMID 20098110
- [Background] Yoshimura K, Asano Y, Aoi N, Kurita M, Oshima Y, Sato K, Inoue K, Suga H, Eto H, Kato H, Harii K. Progenitor-enriched adipose tissue transplantation as rescue for breast implant complications. Breast J. 2010 Mar-Apr;16(2):169-75. doi: 10.1111/j.1524-4741.2009.00873.x. Epub 2009 Nov 12. PMID 19912236

RESULTS

PARTICIPANT FLOW:
Groups:
- Fat Grafting: Fat Grafting procedure designed to deliver an autologous fat graft admixed with autologous stromal vascular fraction (SVF) at a high cell dose.
Period: Overall Study
Arm/Group | Fat Grafting
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fat Grafting
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 5
Skin Volume (cc) [Median (Standard Deviation); unit: cc] | 5 (0)
Skin Thickness (mm) [Median (Standard Deviation); unit: mm] | 5 (0)

OUTCOME MEASURES:

1. Primary Outcome: Average Fat Graft Volume Facial Form From Baseline up to 9 Months
Description: High resolution CT scanning with 3D reconstruction at 0, 1, 3, and 9 months
Time Frame: 0, 1, 3, and 9 months
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Fat Grafting
Number analyzed (Participants) | 5
cc
  9 month | 3.46 (3.42)
  3 months | 3.95 (3.77)
  1 months | 5.98 (5.80)
  0 months | 0 (0)

2. Primary Outcome: Average Tissue Thickness From Baseline up to 9 Months
Description: High resolution CT scanning with 3D reconstruction at 0, 1, 3, and 9 months
Time Frame: 0, 1, 3, and 9 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Fat Grafting
Number analyzed (Participants) | 5
mm
  9 month | 13.62 (5.96)
  3 months | 14.1 (5.76)
  1 months | 15.62 (5.89)
  0 months | 11.00 (5.78)

3. Secondary Outcome: Measure Quality of Life in Subjects After Grafting Using Validated Psychosocial Measures.
Description: 1) Social Avoidance and Distress Scale (SADS) uses a questionnaire including 28 true/false items, with scores ranging from 0-10. A "low" score is below 4, "high" is above 7; intermediate is between 4-7. 2) COPE scale asks the subject to indicate what he/she generally does and feels, when he/she experience stressful events. On a scale of 60-240 where the higher ends indicates the subject does this activity most frequently during stressful events; 3) The Satisfaction With Appearance Scale (SWAP) is a 14-item questionnaire, assessing both the subjective appraisal and social-behavioral components of body image, where the higher the score, the more satisfied subject is with procedure, ranging from 0-7 for a total possible score range between 0-98 .
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale, see outcome measure de
Arm/Group | Fat Grafting
Number analyzed (Participants) | 5
units on a scale, see outcome measure de
  SADS Scale | 9.3 (8.1)
  COPE | 67.2 (14.5)
  SWAP | 18.8 (22.1)

4. Secondary Outcome: Composition of SVF
Description: Cell assessment included stromal vascular fraction composition evaluated by flow cytometry.
Time Frame: time of fat grafting, up to 12 hours post-baseline
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Fat Grafting
Number analyzed (Participants) | 5
percentage of cells
  % Endothelial Cells | 9.76 (6.24)
  % Pericytes | 9.91 (5.22)
  % Supradventitial Stromal Cells | 65.5 (12.5)

5. Secondary Outcome: Characterization of Adipose Stromal Cell (ASC) Function
Description: Cell assessment will include viable stromal vascular fraction per gram of lipoaspirate.
Time Frame: time of surgery, up to 12 hours post-baseline
Measure: Mean (Standard Deviation); unit: mL of viable SVF per g of lipoaspirate
Arm/Group | Fat Grafting
Number analyzed (Participants) | 5
mL of viable SVF per g of lipoaspirate | 23.444 (1.924)

ADVERSE EVENTS:
Groups:
- Fat Grafting: Autologous fat grafting is a potential solution. Grafting of autologous fat tissue is a minimally invasive surgical technique that starts with the harvest of fat tissue from the abdomen or thighs using liposuction through incisions less than 5mm in length. The lipoaspirate is then processed to concentrate the adipose fraction and reinjected into the donor site. This surgical procedure involves the immediate transplantation of a patient's own tissue in a single operative procedure. It has the advantages of:
  * Minimal access incisions
  * Ability to transfer significant amounts of tissue (hundreds of grams of tissue)
  * Can be used in setting of previous surgical procedures and presence of hardware
  * Usually performed as outpatient procedure
  * Minimal donor site morbidity at graft harvest site
  * Low risk compared with more invasive surgical procedures
  * Can be repeated multiple times, if necessary, even using the same donor site
Arm/Group | Fat Grafting
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No